CLINICAL TRIAL: NCT05088057
Title: A Phase Ⅱ Study to Evaluate the Efficacy and Safety of Camrelizumab Plus Chemotherapy as Neoadjuvant Therapy With Triple Negative Breast Cancer (TNBC)
Brief Title: Neoadjuvant Camrelizumab Plus Chemotherapy in Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aiping Shi (Other)
Responsible Party: Sponsor-Investigator, Aiping Shi, The First Hospital of Jilin University, Jilin University
Organization: Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-TNBC-01
Record Dates: First submitted 2021-10-11; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Triple Negative Breast Cancer (TNBC)
Keywords: Camrelizumab; Chemotherapy; Neoadjuvant; PD-1
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab; Doxorubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Chemotherapy (Experimental): PD-1+AC-T: Participants receive Camrelizumab Q3W + doxorubicin Q3W + cyclophosphamide Q3W for 4 cycles, followed by Camrelizumab Q3W + docetaxel Q3W for 4 cycles as neoadjuvant therapy prior to surgery,followed by 9 cycles of Camrelizumab Q3W as adjuvant therapy post-surgery.
  PD-1+TA: Participants receive Camrelizumab Q3W for 8 cycles , docetaxel Q3W + doxorubicin Q3W for 4 cycles as neoadjuvant therapy prior to surgery,followed by 9 cycles of Camrelizumab Q3W as adjuvant therapy post-surgery.
  Interventions: Drug: Camrelizumab; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Docetaxel

INTERVENTIONS:
Drug: Camrelizumab — 200mg on Day 1 of each cycle in the neoadjuvant and adjuvant phases of the study for a total of 17 cycles (Q3W), intravenous (IV) infusion.
Drug: Doxorubicin — 60mg/m² on Day 1 of Cycles 1-4 (Q3W)of the neoadjuvant phase of the study, IV infusion.
Drug: Cyclophosphamide — 600 mg/m² on Day 1 of Cycles 1-4 (Q3W)of the neoadjuvant phase of the study, IV infusion.
Drug: Docetaxel — 75mg/m² on Day 1 of Cycles 1-4 (Q3W) or Cycles 5-8 (Q3W) of the neoadjuvant phase of the study, IV infusion;

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Camrelizumab plus chemotherapy as neoadjuvant therapy and Camrelizumab as adjuvant therapy in participants who have triple negative breast cancer (TNBC).

DETAILED DESCRIPTION:
After a screening phase of approximately 28 days, each participant will receive neoadjuvant study treatment (camrelizumab + chemotherapy) for approximately 24 weeks (8 cycles). Each participant will then undergo definitive surgery 2-4 weeks after the last cycle of the neoadjuvant treatment. After definitive surgery, each participant will receive adjuvant study treatment (camrelizumab) for approximately 27 weeks (9 cycles). Following adjuvant study treatment, each participant will be monitored for safety, survival and disease recurrence.

The primary study hypothesis is that camrelizumab is superior to chemotherapy, in combination with chemotherapy, as measured by the rate of Pathological Complete Response (pCR), Event-free Survival (EFS) and Objective Overall Response Rate (ORR) in participants with TNBC.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 Years, female;
2. Histologically documented Triple Negative Breast Cancer (TNBC) patients;
3. The subtypes of TNBC patients should include basal cell-like subtypes (BL1, BL2), Luminal androgenic type (LAR), and other types, such as mesenchymal type (M), mesenchymal stem cell type (MSL) and immunomodulatory type (IM);
4. Previously untreated non-metastatic (M0) TNBC, the primary tumor (T) and regional lymph node (N) combined staging determined by the investigator based on radiological and/or clinical evaluation. Stage at presentation: T1c, N1-N2; T2, N0-N2; T3, N0-N2;
5. Promising radical surgical treatment;
6. At least one measurable lesion according to RECIST 1.1;
7. Life expectancy is not less than 3 months;
8. ECOG: 0～1;
9. Adequate function of major organs meets the following requirements:

   Neutrophils ≥ 1.5×10^9/L Hemoglobin ≥ 90g/L Platelets ≥ 100×10^9/L Total bilirubin≤ 1.5 × the upper limit of normal (ULN) ALT and AST ≤ 2.5 × ULN Serum creatinine ≤1.5 × ULN, Endogenous creatinine clearance ≥50mL/min;
10. Left ventricular ejection fraction (LVEF) ≥50% or ≥ limit of normal (LLN) was evaluated by echocardiography (ECHO) or Multigated Acquisition (MUGA);
11. Women with childbearing potential who are must agree to take effective contraceptive measures during the study period and ≥120 days after the last administration of the study drug, and must have a negative serum pregnancy test result within 7 days prior to initiation of study drug.
12. The patient voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with follow-up;

Exclusion Criteria:

1. Has participated in an interventional clinical study with an investigational compound within 4 weeks prior to initiation of study treatment;
2. Prior treatment with anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4), anti-programmed death-1 (anti-PD-1), and anti-PD-L1 therapeutic antibodies;
3. Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer;
4. Active or history of autoimmune disease or immune deficiency diseases except history of autoimmune-related hypothyroidism, controlled Type 1 diabetes mellitus;;
5. Has a history of (non-infectious) pneumonitis, interstitial lung disease or uncontrollable systematicness diseases, including pulmonary fibrosis, acute lung disease, etc.;
6. Administration of a live attenuated vaccine within 30 days prior to initiation of study treatment or anticipation of need for such a vaccine during the study;
7. Has active infection (CTCAE≥2) needed the treatment of antibiotic within 2 weeks prior to initiation of study treatment;
8. Has a history of serious cardiovascular disease, including myocardial infarction, acute coronary syndrome or coronary angioplasty/stent implantation/bypass grafting history in the past 6 months, and have level II-IV congestion Heart failure (CHF), or III NYHA and IV CHF history;
9. Prior allogeneic stem cell or solid organ transplantation
10. History of neurological or psychiatric disorders, including schizophrenia, severe depressive disorder, bipolar disorder, etc.;
11. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
12. History of severe hypersensitivity reactions to other monoclonal antibodies, or intravenous infusion, or Doxorubicin, or cyclophosphamide, or docetaxel;
13. Female patients during pregnancy and lactation, fertile women with positive baseline pregnancy tests or women of childbearing age who are unwilling to take effective contraceptive measures throughout the trial;
14. Any other situation evaluated by researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-08-19 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | Up to approximately 12-30 weeks
  pCR rate is defined as the percentage of participants without invasive cancer in the breast irrespective of ductal carcinoma in situ or nodal involvement following completion of neoadjuvant systemic therapy by current AJCC staging criteria assessed by the local pathologist at the time of definitive surgery in all participants

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | Up to approximately 2 years
  EFS is defined as the time from start of study treatment to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Objective Overall Response Rate (ORR) | [Time Frame: Up to approximately 12-30 weeks]
  ORR was defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until definitive surgery or disease progression.
Overall survival (OS) | Up to approximately 2 years
  OS is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the analysis will be censored at the date of the last follow-up.
Adverse events (AEs) | Up to approximately 35 weeks
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0. In general, AEs are graded according to the following: Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE. The type, grade and frequency of AEs will be reported.

OTHER OUTCOMES:
End point of exploratory study | Up to approximately 35 weeks
  Correlation analysis and COX regression analysis were performed on pCR, EFS, ORR, OS of patients with basal cell-like subtypes (BL1, BL2), Luminal androgenic type (LAR), and other types.

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Shi, PhD, Study Director — The First Hospital of Jilin University
Locations (1):
- Aiping Shi, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No